CLINICAL TRIAL: NCT03618511
Title: Interventions to Improve HIV Antiretroviral Therapy Adherence in Sofala Province Mozambique
Brief Title: Interventions to Improve HIV Antiretroviral Therapy Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Beira Operational Research Center (Unknown)
Responsible Party: Principal Investigator, James Riddell, Clinical Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00133179
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Financial Incentive Group (Experimental)
  Interventions: Behavioral: Financial Incentive
- Reminders Group (Experimental)
  Interventions: Behavioral: Reminders
- Financial Incentive and Reminders Group (Experimental)
  Interventions: Behavioral: Financial Incentive and Reminders
- Control Group (No Intervention)
- Information Group (Experimental)
  Interventions: Behavioral: Information
- Stigma-relieving Group (Experimental)
  Interventions: Behavioral: Stigma-relieving
- Information and Stigma-relieving Group (Experimental)
  Interventions: Behavioral: Information and Stigma-relieving

INTERVENTIONS:
Behavioral: Financial Incentive — Financial Incentive: Participants will receive monthly financial incentives each time they refill the ART medication on time for six months
  Arms: Financial Incentive Group
Behavioral: Reminders — Reminders: Participants will receive monthly reminder phone calls before their ART medication refill is due for six months.
  Arms: Reminders Group
Behavioral: Financial Incentive and Reminders — Interaction: Participants receive both the Financial Incentives and Reminder Calls.
  Arms: Financial Incentive and Reminders Group
Behavioral: Information — Information: show the participants a video about HIV progression, mechanism of ART, the benefit of adhering to ART.
  Arms: Information Group
Behavioral: Stigma-relieving — Stigma-Reliving: Upon recruitment, inform the participants of the results of a recent population survey regarding people's attitudes towards HIV, if they overestimate the social stigma related to HIV. This intervention intends to reduce the stigma-concern faced by the patients.
  Arms: Stigma-relieving Group
Behavioral: Information and Stigma-relieving — Information and Stigma-relieving: Upon recruitment, show the participants a video about HIV progression, mechanism of ART, the benefit of adhering to ART. In addition, inform the participants of the results of a recent population survey regarding people's attitudes towards HIV, if they overestimate the social stigma related to HIV. This intervention intends to reduce the stigma-concern faced by the patients.
  Arms: Information and Stigma-relieving Group

SUMMARY:
This study will explore whether financial incentives, reminders, information about HIV/AIDS and its treatment and anti-stigma counseling help improve anti-retroviral therapy (ART) adherence among HIV infected individuals in a resource-limited environment. The interventions will be randomized in the study population in a cross-cutting design, with a control group, a financial incentive treatment group, a reminders treatment group, a treatment group that receives both the financial incentive and reminder interventions. In addition, there will be an information treatment group, a stigma-relieving treatment group and a group that receives both information and stigma-relieving interventions. The primary outcomes of interest for this study will be the adherence to ART, measured by attendance rates at clinic appointments and refill collection rates.

ELIGIBILITY:
Inclusion Criteria:

* Infected with HIV;
* Have not start ART, or started ART less than 90 days before;
* Have a phone number on which can discuss private health matters.

Exclusion Criteria:

* Not infected with HIV;
* On ART for more than 90 days;
* Do not have a private phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Medication possession ratio (MPR) at least 95%, 6 month window | 0-6 month interval from date of study enrollment
  Fraction of participants for whom MPR is greater than or equal to 95%. MPR is proportion of days that a respondent is in possession of at least one ART dose. MPR is computed from pharmacy dispensing records. Measurement window truncated to last visit date for patients who transfer clinics, opt out of future study participation, or die.

SECONDARY OUTCOMES:
Medication possession ratio (MPR) at least 95%, 3 month window | 0-3 month interval from date of study enrollment
  Fraction of participants for whom MPR is greater than or equal to 95%. MPR is proportion of days that a respondent is in possession of at least one ART dose. MPR is computed from pharmacy dispensing records. Measurement window truncated to last visit date for patients who transfer clinics, opt out of future study participation, or die.
Medication possession ratio (MPR) at least 80%, 6 month window | 0-6 month interval from date of study enrollment
  Fraction of participants for whom MPR is greater than or equal to 80%. MPR is proportion of days that a respondent is in possession of at least one ART dose. MPR is computed from pharmacy dispensing records. Measurement window truncated to last visit date for patients who transfer clinics, opt out of future study participation, or die.
Medication possession ratio (MPR) at least 80%, 3 month window | 0-3 month interval from date of study enrollment
  Fraction of participants for whom MPR is greater than or equal to 80%. MPR is proportion of days that a respondent is in possession of at least one ART dose. MPR is computed from pharmacy dispensing records. Measurement window truncated to last visit date for patients who transfer clinics, opt out of future study participation, or die.
Appointment attendance rate (AAR) | 0-6 month interval from date of study enrollment
  Average AAR among participants. AAR is proportion of scheduled visits completed during the observation period. "Completed visit" considered done if patient visits clinic on scheduled appointment date, or up to 7 days prior to that date. AAR is computed from clinic records. Measurement window truncated to last visit date for patients who transfer clinics, opt out of future study participation, or die.
Lost to follow-up (LTFU) | 0-6 month interval from date of study enrollment
  Fraction of participants lost to follow up (LTFU). LTFU indicates patient missed last appointment and 90 or more days have elapsed since patient's last scheduled appointment date, with no clinic record of contact since that date. Patients who transfer clinics or opt out of future study participation are excluded from LTFU denominator, but those who die are retained in LTFU denominator.
Test Referral, 1-month window | 1 month interval from date of study enrollment
  This is a binary variable, which takes value 1 if the participant has a successful referral to test for HIV within 1 month of recruitment and 0 otherwise. A participant is considered having a successful referral if someone approaches our study team in the clinic, present us with the proof of an HIV testing together with the barcode-card we distributed to the participant upon recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: James Riddell IV, MD, Principal Investigator — University of Michigan
Locations (1):
- Munhava Health Center, Beira, Sofala, Mozambique

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT03618511/SAP_000.pdf